CLINICAL TRIAL: NCT06471686
Title: Safety of Acamprosate in Treating Alcohol Use Disorder in the Post Liver Transplant Populations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Hyosun Han, Assistant Professor of Clinical medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-19-00991
Record Dates: First submitted 2024-06-10; First posted 2024-06-24 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder; Liver Transplant; Complications
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acamprosate (Experimental): The intervention group was assigned to acamprosate 666 mg oral tablets three times daily in addition to routine medical care for 14 weeks. Once assigned to this group, participants underwent a medication reconciliation with a transplant pharmacist to ensure there were no drug-drug interactions and answer questions regarding the medication. The medication prescription was then sent by the principal investigator (HH) to the patient preferred pharmacy. The research assistants (KL and JA) would confirm that the medication was obtained. They then underwent weekly telemedicine visits with a research member for 14 weeks and filled out self-report surveys to evaluate cravings, alcohol use, and side effects
  Interventions: Drug: Acamprosate
- Standard of Care (No Intervention): The control group continued with what was considered routine medical care as indicated by their medical condition including frequency of clinic visits (ranging from 1-6 months dependent on time from transplant), frequency of laboratory draws (ranging from twice monthly to biannually dependent on time from transplant), and adjustment of LT related medications (i.e. immunosuppression and prophylaxis against communicable disease). They also underwent weekly telemedicine visits with a research member for 14 weeks and filled out self-report surveys to evaluate cravings, alcohol use, and side effects

INTERVENTIONS:
Drug: Acamprosate — 2 pills three times a day
  Other Names: acamprosate pills
  Arms: Acamprosate

SUMMARY:
Acamprosate for alcohol use disorder may benefit liver transplant (LT) recipients with alcohol-associated liver disease (ALD), yet data on feasibility and safety in LT recipients are lacking. This was a single-center unblinded randomized controlled trial of adults (≥18 years) with LT for ALD enrolled between 2021-2023 who were randomized 2:1 to the intervention of acamprosate (666mg dose three time daily) or standard of care (SOC) for 14 weeks. The primary outcome was safety [prevalence of adverse events (AE)]. Secondary outcomes included feasibility (weekly survey response rate >60%), adherence (self reported acamprosate use>60%), and efficacy (reduction in Penn Alcohol Craving Scale [PACS]) and relapse). Relapse was defined as blood phosphatidylethanol≥20ng/mL or reported alcohol use. All analyses were done in the intention to treat (ITT) population and per-protocol population (PPP) (excluding withdrawals/acamprosate non-adherent).

DETAILED DESCRIPTION:
Acamprosate for alcohol use disorder may benefit liver transplant (LT) recipients with alcohol-associated liver disease (ALD), yet data on feasibility and safety in LT recipients are lacking.

This was a single-center unblinded randomized controlled trial of adults (≥18 years) with LT for ALD enrolled between 2021-2023 who were randomized 2:1 to the intervention of acamprosate (666mg dose three time daily) or standard of care (SOC) for 14 weeks. The primary outcome was safety [prevalence of adverse events (AE)]. Secondary outcomes included feasibility (weekly survey response rate >60%), adherence (self reported acamprosate use>60%), and efficacy (reduction in Penn Alcohol Craving Scale [PACS]) and relapse). Relapse was defined as blood phosphatidylethanol≥20ng/mL or reported alcohol use. All analyses were done in the intention to treat (ITT) population and per-protocol population (PPP) (excluding withdrawals/acamprosate non-adherent).

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* must have received a transplant for liver disease secondary to alcohol-associated hepatitis or alcohol-associated cirrhosis
* greater than 24 hours of abstinence.

Exclusion Criteria:

* patients with hypersensitivity to acamprosate calcium or any of its components
* severe renal impairment (creatinine clearance ≤30 mL/min)
* substance dependence other than THC, alcohol, or nicotine
* need for inpatient detoxification or inpatient treatment of alcohol use
* participation in a clinical trial within the past 60 days
* women of childbearing potential without a medically acceptable form of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 14 weeks
  prevalence of adverse events (AE) by common toxicity criteria
Incidence of Treatment-Emergent Liver Test Changes | 14 weeks
  prevalence of liver test abnormalities [aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), total bilirubin

SECONDARY OUTCOMES:
Proportion of participants with weekly survey response rate >60% | 14 weeks
  Feasibility was defined as a response rate >60% to weekly surveys in both treatment groups
Rate of acamprosate usage> 60% | 14 weeks
  Adherence to acamprosate was measured via self-reported total milligrams of acamprosate taken weekly. Participants were deemed adherent to acamprosate to if they utilized it as prescribed for ≥60% of weeks (9 of 14 weeks).
Change in alcohol cravings | 14 weeks
  Cravings were assessed using the validated survey Penn Alcohol Craving Scale . This is a 5 item Likert scale to measure cravings to drink alcohol within the past week with total scores ranging from 0-30. PACS scores were summarized in 4-week increments with the highest PACS score within +/- 2 weeks reported when missing at the specific time point. The median change in baseline PACS score was utilized in the analysis.
change in alcohol use | 14 weeks
  Alcohol use was assessed using a modified Timeline Followback (TFLB) which is a calendar-based method to examine variability, pattern, and extent of drinking using dates to enhance recall within the past 90 days prior to enrollment at baseline and then weekly thereafter until completion of the study. number of standard alcohol drinks per day were calculated based upon the above data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Background] Cholankeril G, Ahmed A. Alcoholic Liver Disease Replaces Hepatitis C Virus Infection as the Leading Indication for Liver Transplantation in the United States. Clin Gastroenterol Hepatol. 2018 Aug;16(8):1356-1358. doi: 10.1016/j.cgh.2017.11.045. Epub 2017 Dec 1. No abstract available. PMID 29199144
- [Background] Ilyas F, Ali H, Patel P, Basuli D, Giammarino A, Satapathy SK. Rising alcohol-associated liver disease-related mortality rates in the United States from 1999 to 2022. Hepatol Commun. 2023 Jun 14;7(7):e00180. doi: 10.1097/HC9.0000000000000180. eCollection 2023 Jul 1. PMID 37314743
- [Background] Cotter TG, Sandikci B, Paul S, Gampa A, Wang J, Te H, Pillai A, Reddy KG, di Sabato D, Little EC, Sundaram V, Fung J, Lucey MR, Charlton M. Liver transplantation for alcoholic hepatitis in the United States: Excellent outcomes with profound temporal and geographic variation in frequency. Am J Transplant. 2021 Mar;21(3):1039-1055. doi: 10.1111/ajt.16143. Epub 2020 Aug 13. PMID 32531107
- [Background] Heyes CM, Schofield T, Gribble R, Day CA, Haber PS. Reluctance to Accept Alcohol Treatment by Alcoholic Liver Disease Transplant Patients: A Qualitative Study. Transplant Direct. 2016 Sep 7;2(10):e104. doi: 10.1097/TXD.0000000000000617. eCollection 2016 Oct. PMID 27795986
- [Background] DiMartini A, Dew MA, Day N, Fitzgerald MG, Jones BL, deVera ME, Fontes P. Trajectories of alcohol consumption following liver transplantation. Am J Transplant. 2010 Oct;10(10):2305-12. doi: 10.1111/j.1600-6143.2010.03232.x. Epub 2010 Aug 19. PMID 20726963
- [Background] Yoo ER, Cholankeril G, Ahmed A. Treating Alcohol Use Disorder in Chronic Liver Disease. Clin Liver Dis (Hoboken). 2020 Mar 26;15(2):77-80. doi: 10.1002/cld.881. eCollection 2020 Feb. PMID 32226621
- [Background] Rabiee A, Mahmud N, Falker C, Garcia-Tsao G, Taddei T, Kaplan DE. Medications for alcohol use disorder improve survival in patients with hazardous drinking and alcohol-associated cirrhosis. Hepatol Commun. 2023 Mar 24;7(4):e0093. doi: 10.1097/HC9.0000000000000093. eCollection 2023 Apr 1. PMID 36972386
- [Background] Ayyala D, Bottyan T, Tien C, Pimienta M, Yoo J, Stager K, Gonzalez JL, Stolz A, Dodge JL, Terrault NA, Han H. Naltrexone for alcohol use disorder: Hepatic safety in patients with and without liver disease. Hepatol Commun. 2022 Dec;6(12):3433-3442. doi: 10.1002/hep4.2080. Epub 2022 Oct 25. PMID 36281979
- [Background] Weinrieb RM, Van Horn DH, McLellan AT, Alterman AI, Calarco JS, O'Brien CP, Lucey MR. Alcoholism treatment after liver transplantation: lessons learned from a clinical trial that failed. Psychosomatics. 2001 Mar-Apr;42(2):110-6. doi: 10.1176/appi.psy.42.2.110. PMID 11239123
- [Background] Rogal S, Youk A, Zhang H, Gellad WF, Fine MJ, Good CB, Chartier M, DiMartini A, Morgan T, Bataller R, Kraemer KL. Impact of Alcohol Use Disorder Treatment on Clinical Outcomes Among Patients With Cirrhosis. Hepatology. 2020 Jun;71(6):2080-2092. doi: 10.1002/hep.31042. Epub 2020 May 22. PMID 31758811
- [Background] Im GY, Mellinger JL, Winters A, Aby ES, Lominadze Z, Rice J, Lucey MR, Arab JP, Goel A, Jophlin LL, Sherman CB, Parker R, Chen PH, Devuni D, Sidhu S, Dunn W, Szabo G, Singal AK, Shah VH. Provider Attitudes and Practices for Alcohol Screening, Treatment, and Education in Patients With Liver Disease: A Survey From the American Association for the Study of Liver Diseases Alcohol-Associated Liver Disease Special Interest Group. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2407-2416.e8. doi: 10.1016/j.cgh.2020.10.026. Epub 2020 Oct 16. PMID 33069880
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Rief W, Barsky AJ, Glombiewski JA, Nestoriuc Y, Glaesmer H, Braehler E. Assessing general side effects in clinical trials: reference data from the general population. Pharmacoepidemiol Drug Saf. 2011 Apr;20(4):405-15. doi: 10.1002/pds.2067. Epub 2010 Nov 8. PMID 21442687
- [Background] Robinson SM, Sobell LC, Sobell MB, Leo GI. Reliability of the Timeline Followback for cocaine, cannabis, and cigarette use. Psychol Addict Behav. 2014 Mar;28(1):154-62. doi: 10.1037/a0030992. Epub 2012 Dec 31. PMID 23276315
- [Derived] Ayyala-Somayajula D, Bottyan T, Shaikh S, Lee BP, Cho SH, Dodge JL, Terrault NA, Han H. Safety of acamprosate for alcohol use disorder after liver transplant: A pilot randomized controlled trial. Liver Transpl. 2025 Apr 1;31(4):498-507. doi: 10.1097/LVT.0000000000000475. Epub 2024 Sep 3. PMID 39225670

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT06471686/Prot_SAP_ICF_000.pdf